CLINICAL TRIAL: NCT06006611
Title: Risk Factors for Severe Disease in Hospitalized Patients With COVID-19 and the Effect
Brief Title: Risk Factors for Severe Disease in Hospitalized Patients With COVID-19 and the Effect of Azvudine Treatment: a Retrospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.BAS.001
Record Dates: First submitted 2023-08-21; First posted 2023-08-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19; Azvudine; severity
MeSH Terms: conditions — COVID-19 | interventions — azvudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Azvudine group: Azvudine group included COVID-19 patients treated with azvudine antiviral therapy;
  Interventions: Drug: Azvudine
- No antiviral group: No antiviral group included COVID-19 patients treated with no antiviral therapy;
- Monotamivir: Monotamivir group included COVID-19 patients treated with monotamivir antiviral therapy

INTERVENTIONS:
Drug: Azvudine — Received antiviral treatment with azvudine
  Groups: Azvudine group

SUMMARY:
The purpose of this study is to explore the factors that can affect the development of severe cases in hospitalized patients with COVID-19, including basic diseases, laboratory parameters, and clinical manifestations; In addition,to explore whether Azvudine can reduce the mortality of hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
4201 COVID-19 patients discharged from our hospital were enrolled. Binary logistic regression analysis and ROC curve were used to investigate the role of comorbidities, laboratory parameters and clinical manifestation on progression of COVID-19 patients. We used propensity-score models conditional on baseline characteristics and Univariate Cox regression model to examine whether Azvudine can reduce the mortality of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

The COVID-19 positive patients

Exclusion Criteria:

1. patients treated with both azvudine and monotamivir;
2. patients receiving other antiviral drugs such as nematavir/ritonavir;
3. age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The COVID-19 positive patients
Sampling Method: Non-Probability Sample
Enrollment: 4201 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality of COVID-19 patients | Time from onset to death
  All-cause mortality of COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Publication of academic papers